CLINICAL TRIAL: NCT03755765
Title: Exploratory Pilot Studies to Demonstrate Mechanisms of Preventing Antibiotic-Associated Diarrhea and the Role for Probiotics
Brief Title: Mechanisms of Preventing Antibiotic-Associated Diarrhea and the Role for Probiotics
Acronym: YOBIOTIC
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Georgetown University (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH); University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Daniel Merenstein, Director of Research Programs, Georgetown University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 2018-0736; 1R61AT009622-01A1 (NIH)
Record Dates: First submitted 2018-11-18; First posted 2018-11-28 (Actual); Results first posted 2023-02-17 (Actual); Last update posted 2023-02-17 (Actual); Status verified 2023-02

CONDITIONS: Antibiotic-associated Diarrhea
MeSH Terms: interventions — Amoxicillin-Potassium Clavulanate Combination

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Control (Placebo Comparator): Yogurt without Bifidobacterium animalis subsp. lactis BB-12 (BB-12) and Amoxicillin-Clavulanate 875 Mg-125 Mg Oral Tablet
  Interventions: Drug: Amoxicillin-Clavulanate 875 Mg-125 Mg Oral Tablet; Other: Control
- BB-12 (Experimental): Bifidobacterium animalis subsp. lactis BB-12 (BB-12)-supplemented yogurt and Amoxicillin-Clavulanate 875 Mg-125 Mg Oral Tablet
  Interventions: Drug: Amoxicillin-Clavulanate 875 Mg-125 Mg Oral Tablet; Biological: BB-12

INTERVENTIONS:
Drug: Amoxicillin-Clavulanate 875 Mg-125 Mg Oral Tablet — Amoxicillin-Clavulanate 875 Mg-125 Mg Oral Tablet
  Other Names: Augmentin
Biological: BB-12 — Bifidobacterium animalis subsp. lactis BB-12-supplemented yogurt
  Arms: BB-12
Other: Control — Yogurt without Bifidobacterium animalis subsp. lactis BB-12 (BB-12)
  Arms: Control

SUMMARY:
The focus of the study is to better understand the mechanisms causing antibiotic-associated diarrhea (AAD) and how probiotics may prevent some of the iatrogenic effects of antibiotic medications. One of the most common indications for probiotics is for prevention of antibiotic-associated diarrhea. Clinically, different probiotic strains have demonstrated the ability to prevent AAD; however, the mechanism of action behind this effect has not been elucidated. Data from several studies suggest that antibiotic-induced disruption of commensal bacteria in the colon results in a significant (up to 50%) reduction in short chain fatty acid (SCFA) production and a concomitant reduction in Na-dependent fluid absorption resulting in AAD. Probiotics have been shown to ameliorate a variety of gastrointestinal disease states and thus, the study investigators hypothesize that administration of a probiotic yogurt will protect against the development of AAD.

DETAILED DESCRIPTION:
Probiotics are live microorganisms that, when administered in adequate amounts, confer a health benefit on the host. One of the most common indications for probiotic treatment is the prevention of antibiotic-associated diarrhea (AAD). Unfortunately, the efficacy of many probiotic products used for AAD is not supported by rigorous independent research, and non-evidence-based clinical usage is common. Data from several studies are consistent with the notion that antibiotic-induced disruption of commensal bacteria in the colon results in a significant reduction of short chain fatty acid (SCFA) production and a concomitant reduction in Na-dependent fluid absorption resulting in AAD. The probiotic strain being studied, Bifidobacterium animalis subsp. lactis BB-12 (BB-12), has been shown to ameliorate a variety of gastrointestinal disease states and is known to produce acetate at concentrations up to 50 mM in vitro. Thus, the investigators hypothesize that administration of BB-12 at the same time as antibiotic consumption will protect against the development of AAD through its ability to generate acetate directly, and also increase other SCFAs through cross-feeding of certain bacteria in the Firmicutes phylum such Clostridium, Eubacterium and Roseburia, which use acetate to produce butyrate.

The primary aim of the R61 phase (N=60) is to determine the ability of BB-12 to impact antibiotic-induced reduction in SCFA as reflected by the levels of acetate, the most abundant primary colonic SCFA. The primary hypothesis is that antibiotics will result in a reduction in fecal SCFA, but BB-12 supplementation will protect against antibiotic-induced SCFA reduction and/or be associated with a more rapid return to baseline SCFA levels as compared to controls. Antibiotics also result in a decrease in total microbial counts and diversity in the gut microbiota, disrupting the homeostasis of the gut ecosystem and allowing colonization by pathogens. The secondary aim will be to determine the ability of BB-12 to impact antibiotic-induced disruption of the gut microbiota with 16S (16 Svedberg) ribosomal ribonucleic acid (rRNA) profiling. The secondary hypothesis is that antibiotics will result in a decrease in the overall number and diversity of bacterial species present in the fecal microbiota, and further BB-12 supplementation will protect against antibiotic-induced shifts in the microbiota and/or will be associated with a more rapid return to a baseline microbiota composition as compared to controls. The long-term goal is to determine the impact of BB-12 on a variety of gastrointestinal disease states and ages, through high-level independent research. This mechanism elucidation is important for directing future translational and effectiveness research.

ELIGIBILITY:
Inclusion Criteria:

1. Has the ability to read, speak, and write in English
2. Has refrigerator (for proper storage of the study yogurt)
3. Has reliable telephone access
4. Is between ages of 18-65 years
5. Agree to refrain from eating yogurts, yogurt drinks, and other foods specified in the provided What Not to Eat list
6. Agree to collect stool samples and participate in follow-up calls as specified

Exclusion Criteria:

1. Diabetes or asthma that requires medication
2. Allergy to strawberry
3. Active diarrhea (three or more loose stools per day for two consecutive days)
4. Any gastrointestinal (or digestive tract) medications, i.e. medicines for irritable bowel syndrome, gastroesophageal (acid) reflux disease, inflammatory bowel disease, etc.
5. History of heart disease, including valvulopathies or cardiac surgery, any implantable device or prosthetic
6. History of gastrointestinal surgery or disease
7. Lactose intolerance that prevents participant from eating yogurt
8. Allergy to milk-protein
9. Allergy to any component of the product or the yogurt vehicle
10. Allergy to penicillin or cephalosporin class antibiotics
11. Allergy to any of the following medications: a) Penicillin; b) Erythromycin; c) Tetracycline; d) Trimethoprim; e) Ciprofloxacin
12. Women who are breastfeeding, pregnant, or planning to become pregnant during the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2019-07-23 (Actual); Primary Completion 2020-01-08 (Actual); Study Completion 2020-01-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Merenstein, MD, Principal Investigator — Georgetown University; Claire Fraser, PhD, Principal Investigator — University of Maryland, Baltimore
Locations (1):
- Georgetown University Department of Family Medicine, Washington D.C., District of Columbia, United States

REFERENCES:
- [Result] Merenstein D, Fraser CM, Roberts RF, Liu T, Grant-Beurmann S, Tan TP, Smith KH, Cronin T, Martin OA, Sanders ME, Lucan SC, Kane MA. Bifidobacterium animalis subsp. lactis BB-12 Protects against Antibiotic-Induced Functional and Compositional Changes in Human Fecal Microbiome. Nutrients. 2021 Aug 17;13(8):2814. doi: 10.3390/nu13082814. PMID 34444974

RESULTS

PARTICIPANT FLOW:
Groups:
- Not Randomized: Withdrawals prior to randomization
Period: Overall Study
Arm/Group | Control | BB-12 | Not Randomized
Started | 20 | 42 | 4
Completed | 18 | 38 | 0
Not Completed | 2 | 4 | 4
Not completed — Withdrawal by Subject | 2 | 4 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | BB-12 | Not Randomized | Total
Number analyzed (Participants) | 20 | 42 | 4 | 66
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.4 (8.1) | 29.6 (10.3) | 31.8 (21.6) | 29.7 (10.6)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 11 | 23 | 1 | 35
  Male | 9 | 18 | 3 | 30
  Not reported | 0 | 1 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 0 | 4
  Not Hispanic or Latino | 18 | 36 | 4 | 58
  Unknown or Not Reported | 0 | 4 | 0 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 3 | 6 | 3 | 12
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 5 | 8 | 0 | 13
  White | 11 | 28 | 1 | 40
  More than one race | 1 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0
Health insurance status [Count of Participants; unit: Participants]
  Yes | 20 | 41 | 4 | 65
  No | 0 | 1 | 0 | 1
Household smoking [Count of Participants; unit: Participants]
  No | 18 | 40 | 4 | 62
  Yes | 2 | 2 | 0 | 4
Marital status [Count of Participants; unit: Participants]
  Married | 4 | 10 | 0 | 14
  Living with a partner | 2 | 5 | 0 | 7
  Single | 14 | 26 | 3 | 43
  Separated | 0 | 0 | 0 | 0
  Divorced | 0 | 0 | 0 | 0
  Widowed | 0 | 1 | 1 | 2
Annual gross total income [Count of Participants; unit: Participants]
  Less than $15,000 | 1 | 6 | 0 | 7
  $15,000-$29,999 | 1 | 3 | 0 | 4
  $30,000-$49,999 | 1 | 5 | 0 | 6
  $50,000-$74,999 | 1 | 5 | 0 | 6
  $75,000-$99,999 | 5 | 6 | 0 | 11
  $100,000-$150,999 | 2 | 2 | 0 | 4
  $150,000-$200,000 | 1 | 1 | 0 | 2
  More than $200,000 | 2 | 6 | 3 | 11
  Prefer not to answer | 0 | 3 | 0 | 3
  Unknown/Not Reported | 6 | 5 | 1 | 12

OUTCOME MEASURES:

1. Primary Outcome: Level of Fecal Short-chain Fatty Acid (SCFA) Acetate
Description: Level of fecal short-chain fatty acid acetate (SCFA) after administration of amoxicillin clavulanate
Time Frame: day 0 (post run-in), 7, 14, 21, 30
Population: Number of samples received
Measure: Mean (Standard Deviation); unit: micromolar (μM)
Arm/Group | Control | BB-12
Number analyzed (Participants) | 12 | 29
micromolar (μM)
  Day 0 | 53.1 (18.0) | 45.2 (20.3)
  Day 7: number analyzed (Participants) | 12 | 27
  Day 7 | 42.3 (17.5) | 38.1 (17.6)
  Day 14 | 36.8 (11.1) | 40.8 (16.1)
  Day 21 | 43.8 (17.6) | 50.5 (20.9)
  Day 30: number analyzed (Participants) | 10 | 26
  Day 30 | 39.8 (14.3) | 44.5 (14.1)

2. Secondary Outcome: Level of Fecal SCFA Propionate
Description: Level of fecal short-chain fatty acid propionate after administration of amoxicillin clavulanate
Time Frame: day 0 (post run-in), 7, 14, 21, 30
Population: Number of samples received
Measure: Mean (Standard Deviation); unit: μM
Arm/Group | Control | BB-12
Number analyzed (Participants) | 12 | 29
μM
  Day 0 | 14.3 (9.1) | 13.0 (7.2)
  Day 7: number analyzed (Participants) | 12 | 25
  Day 7 | 14.3 (6.7) | 12.5 (6.0)
  Day 14 | 11.8 (6.9) | 12.0 (6.1)
  Day 21: number analyzed (Participants) | 11 | 29
  Day 21 | 11.0 (3.5) | 14.8 (7.8)
  Day 30: number analyzed (Participants) | 11 | 26
  Day 30 | 11.4 (7.3) | 11.5 (5.7)

3. Secondary Outcome: Level of Fecal SCFA Butyrate
Description: Level of fecal short-chain fatty acid butyrate (μM) after administration of amoxicillin clavulanate
Time Frame: day 0 (post run-in), 7, 14, 21, 30
Population: Number of samples received
Measure: Mean (Standard Deviation); unit: μM
Arm/Group | Control | BB-12
Number analyzed (Participants) | 12 | 29
μM
  Day 0: number analyzed (Participants) | 11 | 29
  Day 0 | 12.7 (6.2) | 12.7 (8.4)
  Day 7: number analyzed (Participants) | 11 | 24
  Day 7 | 9.0 (5.3) | 8.3 (5.7)
  Day 14 | 7.4 (4.3) | 8.9 (6.1)
  Day 21: number analyzed (Participants) | 11 | 29
  Day 21 | 11.6 (9.2) | 11.9 (7.8)
  Day 30: number analyzed (Participants) | 11 | 26
  Day 30 | 8.3 (5.3) | 9.9 (4.0)

4. Other Pre Specified Outcome: Change in Community Diversity (Shannon Diversity Index) From Pre run-in Baseline
Description: The Shannon diversity metric is a measure of community diversity and takes into account species richness (number of distinct taxa) and the relative abundance of each taxon. The Shannon diversity index was calculated for samples at each time point from subjects receiving control or BB-12 yogurt. The first of two baseline samples was collected from each subject at the time of enrollment (pre run-in) before a 30-day run-in period in which the consumption of dietary probiotics was stopped. A higher index indicates more diversity and a lower index indicates less diversity.
Time Frame: day 0 (pre run-in), 7, 14, 21, 30
Population: Number of samples received
Measure: Mean (Standard Deviation); unit: Shannon Diversity Index
Arm/Group | Control | BB-12
Number analyzed (Participants) | 18 | 38
Shannon Diversity Index
  Day 0 Pre run-in: number analyzed (Participants) | 15 | 31
  Day 0 Pre run-in | 3.711 (0.349) | 3.774 (0.302)
  Day 7: number analyzed (Participants) | 10 | 28
  Day 7 | 3.380 (0.364) | 3.567 (0.479)
  Day 14: number analyzed (Participants) | 13 | 32
  Day 14 | 3.419 (0.465) | 3.632 (0.307)
  Day 21: number analyzed (Participants) | 10 | 27
  Day 21 | 3.709 (0.322) | 3.708 (0.308)
  Day 30: number analyzed (Participants) | 11 | 27
  Day 30 | 3.395 (0.409) | 3.684 (0.397)

5. Other Pre Specified Outcome: Change in Community Diversity (Shannon Diversity Index) From Post run-in Baseline
Description: The Shannon diversity metric is a measure of community diversity and takes into account species richness (number of distinct taxa) and the relative abundance of each taxon. The Shannon diversity index was calculated for samples at each time point from subjects receiving control or BB-12 yogurt. The second baseline sample was collected from each subject after a 30-day run-in period in which the consumption of dietary probiotics was stopped (post run-in). A higher index indicates more diversity and a lower index indicates less diversity.
Time Frame: day 0 (post run-in), 7, 14, 21, 30
Population: Number of samples received
Measure: Mean (Standard Deviation); unit: Shannon Diversity Index
Arm/Group | Control | BB-12
Number analyzed (Participants) | 18 | 38
Shannon Diversity Index
  Day 0 Post run-in: number analyzed (Participants) | 15 | 29
  Day 0 Post run-in | 3.845 (0.290) | 3.718 (0.261)
  Day 7: number analyzed (Participants) | 11 | 25
  Day 7 | 3.528 (0.396) | 3.606 (0.494)
  Day 14: number analyzed (Participants) | 13 | 26
  Day 14 | 3.496 (0.486) | 3.666 (0.304)
  Day 21: number analyzed (Participants) | 10 | 23
  Day 21 | 3.785 (0.295) | 3.727 (0.278)
  Day 30: number analyzed (Participants) | 11 | 23
  Day 30 | 3.486 (0.444) | 3.712 (0.391)

6. Other Pre Specified Outcome: Bray-Curtis Dissimilarity
Description: Community divergence over time with respect to the baseline sample (post run-in, day 0)
Time Frame: day 0, 7, 14, 21, 30
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Change in Diarrhea/Stool Frequency
Description: Change in diarrhea/stool frequency from baseline
Time Frame: day 7, 14, 21, 30
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Pre-run in baseline to day 30
Arm/Group | Control | BB-12
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/42
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/42
Other Adverse Events (participants affected / at risk) | 15/18 | 25/38
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Control (N=18) | BB-12 (N=38)
Loose stool (Gastrointestinal disorders) | 9 | 14
Diarrhea (Gastrointestinal disorders) | 1 | 1
Constipation (Gastrointestinal disorders) | 3 | 4
Flatulence (Gastrointestinal disorders) | 8 | 8
Lack/Loss of Appetite (General disorders) | 3 | 2
Stomach Pain (Gastrointestinal disorders) | 3 | 1
Rash (General disorders) | 0 | 2
Vomiting (Gastrointestinal disorders) | 0 | 2
Dyspepsia (Gastrointestinal disorders) | 3 | 1
Nausea (General disorders) | 5 | 3
Other (General disorders) | 6 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-05-27): https://cdn.clinicaltrials.gov/large-docs/65/NCT03755765/Prot_SAP_001.pdf
  • Informed Consent Form (2019-06-22): https://cdn.clinicaltrials.gov/large-docs/65/NCT03755765/ICF_000.pdf